CLINICAL TRIAL: NCT05220657
Title: Exploring the Relationship Between the Gut Microbiome Based Metagenomic Signature, Physical Fitness Levels and Metabolic Responses to Exercise: a Pilot Study on 50 Healthy Male Volunteers
Brief Title: Exploring the Relationship Between the Gut Microbiome, Physical Fitness Levels and Metabolic Responses to Exercise
Acronym: EXOMIC
Status: Completed | Type: Observational
Sponsor: University of Rennes 2 (Other)
Collaborators: Nahibu (Unknown)
Responsible Party: Principal Investigator, Frédéric Derbré, Associate Professor, University of Rennes 2
Other Study IDs: 2021-A02496-35
Record Dates: First submitted 2022-01-17; First posted 2022-02-02 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2023-01

CONDITIONS: Elite Cyclists; Elite Soccer Players; Sedentary Behavior
Keywords: Physical activity; Carbohydrates and lipid metabolisms; Gut microbiota; Maximal oxygen consumption
MeSH Terms: conditions — Sedentary Behavior; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Frozen stool suspension
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Low active subjects: No intervention
  Interventions: Diagnostic Test: Maximal incremental exercise test; Diagnostic Test: Submaximal exercise test
- Moderately active subjects: No intervention
  Interventions: Diagnostic Test: Maximal incremental exercise test; Diagnostic Test: Submaximal exercise test
- Elite soccer players: No intervention
  Interventions: Diagnostic Test: Maximal incremental exercise test; Diagnostic Test: Submaximal exercise test
- Elite cyclists: No intervention
  Interventions: Diagnostic Test: Maximal incremental exercise test; Diagnostic Test: Submaximal exercise test

INTERVENTIONS:
Diagnostic Test: Maximal incremental exercise test — Gas exchanges are measured during all the test on ergocycle until oxygen consumption reach its maximum value
Diagnostic Test: Submaximal exercise test — A 25-min submaximal exercise test on ergocycle under fasting condition. Gas exchanges are measured during all the test.

SUMMARY:
Gut microbiota are all microorganisms including bacteria and microscopic eukaryotes that live in the digestive tracts of humans or mammals. During the last decade, some authors highlighted that a link exists between gut microbiota and sport performance. In this project, we hypothesize that gut microbiota is able to adapt to the energy needs of the body, really higher in top-level athletes or considerably lower in inactive individuals. In this context, this clinical study aims to characterize the bacterial metagenome of gut microbiota from populations located in a continuum from sedentary people to top-level athletes with high (i.e. soccer players), even very high energy needs (i.e. cyclists). The finality of this project is thus to determine if it exists some bacterial profile allowing to characterize, even to predict, the energy metabolism of an athlete and so the probability to be performant in competition.

DETAILED DESCRIPTION:
Gut microbiota are all microorganisms including bacteria, archaea and microscopic eukaryotes that live in the digestive tracts of humans or mammals. All these microorganisms live in homeostasis in the gastrointestinal tract and provide a variety of benefits to the host immune system and energy metabolism in a state called eubiosis. On contrary, a state of dysbiosis occurs when the diversity of commensal bacteria is reduced especially in some chronic diseases including obesity, cancer or gastrointestinal diseases. During the last decade, substantial studies highlighted that a link exists between gut microbiota composition and sport performance. Research team especially identified a direct link between gut microbiota and skeletal muscle, a key organ in sport performance (Nay et al. 2019). Using rodent models, They observed that 1) the endurance performance was reduced in mice for which the gut microbiome had been experimentally destructed (Nay et al. 2019), and 2) the reduction of endurance performance was due to lower muscle glycogen levels, a key energy substrate for muscle endurance.

Complementary researches have been conducted in humans to characterize the impact of physical activity on gut microbiota composition and function. A study conducted in large American cohort of 1500 individuals have thus highlighted that the gut microbiota diversity was much more important in individuals performing regular physical activity (3-5 times/week or more) compared to physically inactive people. The few studies conducted in top-level athletes are in accordance with these results. Indeed, it has been demonstrated that international Irish rugby players exhibited a clear higher microbial diversity than inactive and sedentary populations associated to higher production of short-chain fatty acids (SCFA), some key energy substrates produced by commensal bacteria (Clarke et al. 2014; Barton et al. 2018). Conversely, when people are completely physically deconditioned such as astronauts under microgravity or bedridden patients, a clear modification of gut microbiota composition occurs in the gastrointestinal tract (Voorhies and al. 2019). Such differences between top-level athletes, inactive or extremely inactive individuals cannot be only explained to lifestyle, especially diet. Indeed, longitudinal studies have clearly showed that a several weeks training period can increase the gut microbial diversity in humans suggesting an increased capacity of gut microbiota to extract energy from food, especially from dietary fibers (Allen et al. 2018). All together, these data support that the gut microbiota could adapt to the energy needs of the body, really higher in top-level athletes or considerably lower in extremely inactive individuals (e.g. astronauts or bedridden patients). These data also suggest that gut microbiota could punctually inform of the body's metabolic state of an individual.

In this context, this clinical study aims to characterize the bacterial metagenome of gut microbiota from populations located in a continuum from sedentary people to top-level athletes with high (i.e. soccer players), even very high energy needs (i.e. cyclists). The finality of this project is thus to determine if it exists some bacterial profile allowing to characterize, even to predict, the energy metabolism of an athlete and so the probability to be performant in competition.

For this purpose, we will assess the metabolic responses to exercise from different athletic populations (i.e. elite cyclists and soccer players) and non-active of moderately active populations. All the volunteers (n=50) will perform 3 visits in the M2S lab: 1) an inclusion visit including anthropometric measures, dietary and physical activity surveys, and after which the volunteer will leave the lab with a Nahibu kit allowing to send us a fecal sample in the next 7 days, 2) a second visit to perform the incremental cycling test, 3) a last visit to perform metabolic measures in fasted condition in basal and during submaximal exercises. The metabolic parameters measured during these tests (e.g. VO2max, power in aerobic and anaerobic thresholds, maximal carbohydrates and lipids oxidation) will be then related to the metagenomic shotgun data obtained in fecal samples.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 18 and 25 kg/m²
* Non-smoker
* Written informed consent

Exclusion Criteria:

* Cardiovascular risks
* Metabolic diseases (e.g. diabetes)
* Use of antibiotics, anti-fungi or anti-parasites in the last 3 months or during participation in the study
* Use of prebiotics and / or probiotics in the form of supplements in the 7 days preceding the start of the study (greater than or equal to 100000000 Colony Forming Units or organisms per day)
* Taking drug treatment for chronic pain management (paracetamol, vasodilator, homeopathy, aspirin greater than 500 mg per day)
* Simultaneous participation in another research involving the human person or having recently participated in another research for which the exclusion period has not been completed.

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Populations located in a continuum from inactive people to top-level athletes with high (i.e. soccer players) and very high energy needs (i.e. cyclists).
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2022-01-20 (Actual); Primary Completion 2022-10-26 (Actual); Study Completion 2022-11-23 (Actual)

PRIMARY OUTCOMES:
Gut microbiota composition | week 1
  Whole metagenomic sequencing using shotgun approach

SECONDARY OUTCOMES:
Gut microbiota function | Week 1
  Whole metagenomic sequencing using shotgun approach
Short chain fatty acids levels in stools | week 1
  Quantification of gut microbiota metabolites will be performed in frozen stool suspension using Ultra Performance Liquid Chromatography - Mass spectrometry.
Amino acids levels in stools | week 1
  Quantification of gut microbiota metabolites will be performed in frozen stool suspension using Ultra Performance Liquid Chromatography - Mass spectrometry.
Maximal oxygen consumption (VO2max) | Week 2
  Maximal oxygen consumption (ml/min/kg) will be determined during maximal incremental ergocycle test. Gas exchanges will be measured throughout the test.
Lipid oxidation during physical exercise | week 3
  A submaximal ergocyle test will be performed under fasting condition. After 4 min of warm-up (60W), subjects will perform 10 min at 50% VO2max and a second 10 min step at 90% of the anaerobic threshold. Measurements of respiratory gas exchange will be used to estimate the type and amount of substrate oxidized and the amount of energy produced during exercise (kcal/min).
Carbohydrate oxidation during physical exercise | week 3
  A submaximal ergocyle test will be performed under fasting condition. After 4 min of warm-up (60W), subjects will perform 10 min at 50% VO2max and a second 10 min step at 90% of the anaerobic threshold. Measurements of respiratory gas exchange will be used to estimate the type and amount of substrate oxidized and the amount of energy produced during exercise (kcal/min).

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric DERBRÉ, PhD, Principal Investigator — Laboratory of Movement, Sport and health Sciences (M2S)
Locations (1):
- University Rennes 2 - Laboratory "Movement, Sport and health Sciences", Bruz, Brittany Region, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nay K, Jollet M, Goustard B, Baati N, Vernus B, Pontones M, Lefeuvre-Orfila L, Bendavid C, Rue O, Mariadassou M, Bonnieu A, Ollendorff V, Lepage P, Derbre F, Koechlin-Ramonatxo C. Gut bacteria are critical for optimal muscle function: a potential link with glucose homeostasis. Am J Physiol Endocrinol Metab. 2019 Jul 1;317(1):E158-E171. doi: 10.1152/ajpendo.00521.2018. Epub 2019 Apr 30. PMID 31039010
- [Background] Clarke SF, Murphy EF, O'Sullivan O, Lucey AJ, Humphreys M, Hogan A, Hayes P, O'Reilly M, Jeffery IB, Wood-Martin R, Kerins DM, Quigley E, Ross RP, O'Toole PW, Molloy MG, Falvey E, Shanahan F, Cotter PD. Exercise and associated dietary extremes impact on gut microbial diversity. Gut. 2014 Dec;63(12):1913-20. doi: 10.1136/gutjnl-2013-306541. Epub 2014 Jun 9. PMID 25021423
- [Background] Barton W, Penney NC, Cronin O, Garcia-Perez I, Molloy MG, Holmes E, Shanahan F, Cotter PD, O'Sullivan O. The microbiome of professional athletes differs from that of more sedentary subjects in composition and particularly at the functional metabolic level. Gut. 2018 Apr;67(4):625-633. doi: 10.1136/gutjnl-2016-313627. Epub 2017 Mar 30. PMID 28360096
- [Background] Voorhies AA, Mark Ott C, Mehta S, Pierson DL, Crucian BE, Feiveson A, Oubre CM, Torralba M, Moncera K, Zhang Y, Zurek E, Lorenzi HA. Study of the impact of long-duration space missions at the International Space Station on the astronaut microbiome. Sci Rep. 2019 Jul 9;9(1):9911. doi: 10.1038/s41598-019-46303-8. PMID 31289321
- [Background] Allen JM, Mailing LJ, Niemiro GM, Moore R, Cook MD, White BA, Holscher HD, Woods JA. Exercise Alters Gut Microbiota Composition and Function in Lean and Obese Humans. Med Sci Sports Exerc. 2018 Apr;50(4):747-757. doi: 10.1249/MSS.0000000000001495. PMID 29166320